CLINICAL TRIAL: NCT00018356
Title: Physiologic Effects of PRMS & Testosterone in the Debilitated Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sullivan, Dennis - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: AGCG-007-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Muscle Weakness; Muscular Atrophy
Keywords: Aging; nutrition; rehabilitation
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy | interventions — Exercise; Testosterone

ARMS (1):
- 1 (Other)
  Interventions: Procedure: exercise; Drug: testosterone

INTERVENTIONS:
Procedure: exercise
Drug: testosterone

SUMMARY:
This study's primary objective is to determine the independent and combined effects of progressive resistance muscle strength training and testosterone on the development of sustainable improvements in physical function.

ELIGIBILITY:
Inclusion Criteria:

The study will be limited to those patients who are metabolically stable and free of metastatic cancer and limiting end organ disease. Their total serum testosterone must be less than 480 and PSA less than 10.

Exclusion Criteria:

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 1999-01; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Sullivan, MD, Principal Investigator — Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock
Locations (1):
- Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas, United States

REFERENCES:
- [Result] Sullivan DH, Roberson PK, Johnson LE, Bishara O, Evans WJ, Smith ES, Price JA. Effects of muscle strength training and testosterone in frail elderly males. Med Sci Sports Exerc. 2005 Oct;37(10):1664-72. doi: 10.1249/01.mss.0000181840.54860.8b. PMID 16260965